CLINICAL TRIAL: NCT07360470
Title: Anatomical Assessment of Orbital Contents on Imaging
Brief Title: Anatomical Assessment of Orbital Contents on Imaging (EACOI)
Acronym: EACOI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0315 - EACOI
Record Dates: First submitted 2025-06-03; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-01

CONDITIONS: Anatomical Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oculomotor muscles study
- Intraorbital content

SUMMARY:
This is a single-center retrospective study based on existing data. The study focuses on the anatomical content of the orbit, and in particular the anatomy of the oculomotor muscles in the orbit, which are involved in eye movements. There are 6 of these muscles, with the superior, inferior, medial and lateral rectus muscles, and the superior and inferior oblique muscles in each orbit. The study also covers the anatomy of the optic nerve and orbital fat.

Knowledge of the anatomy and biometry of the oculomotor muscles, and of methods for assessing these muscles, has implications for clinical, medical and surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* No opposition to the participation
* Usable imaging test

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the general population who underwent brain imaging (CT or MRI) in the medical imaging department
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intra- and inter-observer reproducibility of oculomotor muscle anatomical criteria in imaging | 1 year.
  Evaluate the reproducibility of different oculomotor muscle measurements, such as volume (mm3), surface (mm2) or two-dimensional measurements (mm). Differences to the mean. Intraclass correlation coefficient (ICC).

SECONDARY OUTCOMES:
Reproducibility of measurements of optic nerve size and orbital fat in imaging | 1 year.
  Evaluate the reproducibility of different measurements to assess the size of the optic nerve (volume (mm3), surface (mm2), two-dimensional measurement (mm) and intra-orbital fat (mm3). Dfference to the mean. Intraclass correlation coefficient (ICC).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided